CLINICAL TRIAL: NCT02772471
Title: Development and Evaluation of the ICP Waveform Tracing Capabilities and Safety of HS-1000 Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HeadSense Medical (Industry)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HS-016
Record Dates: First submitted 2016-05-12; First posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Brain Injuries; Intracranial Hypertension
Keywords: intracranial pressure; noninvasive monitoring
MeSH Terms: conditions — Brain Injuries; Intracranial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HS-1000 recording (Experimental): ICP monitoring will be done in parallel for both HS-1000 and invasive ICP monitoring. HS-1000 ICP monitoring intervals will last at least 30 minutes, continuously depending on the patient's clinical condition.
  Interventions: Device: HS-1000

INTERVENTIONS:
Device: HS-1000

SUMMARY:
Invasive intracranial pressure (ICP) monitoring, using modalities such as parenchymal pressure transducer or external ventricular drain (EVD), provides an ICP waveform that encapsulates valuable diagnostic and monitoring clinical information.

HS-1000 device, a proprietary new non-invasive ICP monitor, is expected to display an ICP waveform safely and accurately with minimal discomfort to patients, compared to standard invasive ICP monitoring procedures used at the participating institutions.

DETAILED DESCRIPTION:
A study will be conducted on 100 patients who undergo invasive ICP measurement due to suspected ICP elevation, regardless to etiology. Each enrolled patient will be monitored with the HS-1000 device and data will be collected throughout the entire procedure. Once the data collection is done, results of the non-invasive measurements will be analyzed accordingly. The end-point of the study is to collect at least half an hour of measurements for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women subjects, aged 18 years old and over at screening visit
* Subjects with neuropathology that the principal investigator considers including in this study.
* Survival expectancy greater than 72 hours
* Subject or legal authorized representative (per local regulation) is able and willing to comply with the requirements of the protocol
* Subject or legal authorized representative (per local regulation) is able to understand and sign written informed consent to participate in the study

Exclusion Criteria:

* Local ear infection
* Known allergy or hypersensitivity to any of the test materials or contraindication to test materials
* For women of childbearing potential: pregnancy (positive pregnancy test) or breast-feeding
* Subjects currently enrolled in or less than 30 days post-participation in other investigational device or drug study(s), or receiving other investigational agent(s)
* Any condition that may jeopardize study participation (e.g., abnormal clinical or laboratory finding) or interpretation of study results, or may impede the ability to obtain informed consent (e.g., mental condition)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of ICP values obtained by the HS device that correlate to ICP using current standards | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Per Kristian Eide, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Levinsky A, Papyan S, Weinberg G, Stadheim T, Eide PK. Non-invasive estimation of static and pulsatile intracranial pressure from transcranial acoustic signals. Med Eng Phys. 2016 May;38(5):477-84. doi: 10.1016/j.medengphy.2016.02.009. Epub 2016 Mar 17. PMID 26997563